CLINICAL TRIAL: NCT00396097
Title: A Four Year Open Label Multi Center Randomized Two Arm Study Of Genotropin In Idiopathic Short Stature Patients: Comparing An Individualized, Target Driven Treatment Regimen To Standard Dosing Of Genotropin
Brief Title: Individualized, Target-Driven Treatment Of Children With Idiopathic Short Stature
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6281280
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Idiopathic Short Stature
Keywords: ISS; human growth hormone
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Standard daily HGH treatment
  Interventions: Drug: Genotropin
- Formula-based (Active Comparator): Formula-based dose regimen
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: Genotropin — Compare daily injections of formula-based HGH treatment to daily injections of standard HGH treatment in subjects with Idiopathic Short Stature over 24 months period followed by an exploratory 24 months period.
  Arms: Standard
Drug: Genotropin — Compare daily injections of formula-based HGH treatment to daily injections of standard HGH treatment in subjects with Idiopathic Short Stature over 24 months period followed by an exploratory 24 months period.
  Arms: Formula-based

SUMMARY:
To demonstrate that an individualized, formula-based Genotropin regimen for children with Idiopathic Short Stature will lead to a targeted height gain (to reach the target of 10th percentile (%), or -1.3 SDS) during 24 months of treatment. The endpoint at 4 years is to explore treatment efficiency over four years of two formula-based dose regimens (sub-arms) compared to standard treatment

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children with bone ages between 3 and 10 years of age for males and 3 and 9 years of age for females
* Naive to Growth Hormone treatment

Exclusion Criteria:

* Abnormal karyotype. Small Gestational Age and Skeletal dysplasia.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2006-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (43):
  - Arkansas Children's Hospital, Little Rock, Alaska
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Pediatric Endocrinology of San Diego Medical Group Incorporated, San Diego, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Memorial Pediatric Specialty Clinic, Colorado Springs, Colorado
  - Pediatric Endocrine Associates, Greenwood Village, Colorado
  - Pediatric Endocrine Associates at The Longmont Clinic, Longmont, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Miller School Of Medicine, University of Miami/Jackson Memorial Medical Center, Miami, Florida
  - Pediatric Endocrinology Associates, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Nancy Wright, MD, Tallahassee, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Johns Hopkins Pediatric Endocrinology, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center Children's Hospital, Springfield, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Endocrine Care of St. Louis, LLC, St Louis, Missouri
  - Saint Barnabas Ambulatory Care Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Women & Children's Hospital of Buffalo, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York (CCMC), Lake Success, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Diabetes & Endocrine Center for Children & Young Adults at Phelps Memorial Hospital, Sleepy Hollow, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Central Ohio Pediatric Endocrinology/Diabetes Services (COPEDS), Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Pediatric Alliance, PC, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Endocrine Clinic P.C., Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Ellen Sher, MD PA, Dallas, Texas
  - Children's Medical Center, Dallas, Texas
  - Cooks Children Medical Center/Dept. of Pediatric Endocrinology, Fort Worth, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281280&StudyName=Individualized%2C%20Target-Driven%20Treatment%20Of%20Children%20With%20Idiopathic%20Short%20Stature

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 4-year, open-label, randomized study conducted at 40 centers across United States of America (USA). The first 2-years of the study constituted core phase and the last 2 years constituted the maintenance phase.
Pre-assignment Details: The participants were randomized in 2:1 manner to formula-based dosing arm and standard dosing arm for initial 2 years of treatment, following which the participants in formula-based dosing arm were re-randomized in a 1:1 manner to one of two physiological doses, for next 2 years, to identify the minimum genotropin dosage to maintain the growth.
Groups:
- Standard Dose Arm: The participants received subcutaneous genotropin, at a maintained standard dose of 0.37 mg/kg/week, throughout the four years.
- Individualized Dose Arm: The participants received subcutaneous genotropin daily, at formula-calculated dose (up to maximum dose of 0.7 mg/kg/week) for the initial 2 years and then lowered to one of two approximately physiological doses (0.18 mg/kg/week or 0.24 mg/kg/week) for the remaining 2 years.
Period: Overall Study
Arm/Group | Standard Dose Arm | Individualized Dose Arm
Started | 114 (4 participants randomized to Individualized Dose, received Standard Dose throughout the study.) | 202
Completed | 88 | 156
Not Completed | 26 | 46
Not completed — Withdrawal by Subject | 17 | 17
Not completed — Lost to Follow-up | 4 | 9
Not completed — Other | 3 | 5
Not completed — Protocol Violation | 0 | 6
Not completed — Adverse Event | 1 | 5
Not completed — Insufficient Clinical Response | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Standard Dose Arm: The participants received subcutaneous genotropin daily, at a maintained standard dose of 0.37 mg/kg/week, throughout the four years.
- Total: Total of all reporting groups
Arm/Group | Standard Dose Arm | Individualized Dose Arm | Total
Number analyzed (Participants) | 114 | 202 | 316
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.3 (2.1) | 8.4 (2.3) | 8.4 (2.2)
Age, Customized [Number; unit: Participants]
  <= 7 years | 37 | 70 | 107
  >=7 years | 77 | 132 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 58 | 89
  Male | 83 | 144 | 227

OUTCOME MEASURES:

1. Primary Outcome: Absolute On-target Difference (AOTD) at 24 Months
Description: This was defined as an absolute difference between the 24-month height standard deviation score (SDS) and targeted 24-month height SDS (10th percentile (%), or -1.3 SDS). SDS indicates how similar the participant was to the reference population. These were calculated using 2000 Center for the Disease Control (CDC) growth reference tables (by age and gender).
Time Frame: 2 years
Population: The Full Analysis Set (FAS) included all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline height SDS value available. Last observation carried forward (LOCF) rule was applied to impute Month 24 missing height SDS data.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Groups:
- Standard Dose Arm: The participants received subcutaneous genotropin daily, at maintained standard dose of 0.37 mg/kg/week, throughout the four years.
Arm/Group | Standard Dose Arm | Individualized Dose Arm
Number analyzed (Participants) | 114 | 202
Standard Deviation Score (SDS) | 0.603 (0.2948) | 0.625 (0.3003)
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm; The null hypothesis was that the individualized treatment arm was not superior to the standard treatment arm; alternative hypothesis that the individualized treatment arm was superior to the standard treatment arm with respect to the mean 24-month AOTD. Using a 2:1 randomization, a two sided sample t-test comparing the root AOTD between the 2 treatment arms with 80% power at a 5% level required 260 subjects. Assuming a 20% attrition rate, approximately 312 subjects were needed for this study; Test type: Superiority or Other; p = 0.5762, ANCOVA; Mean Difference (Final Values) = -0.006, 97.5% CI 1-sided [lower limit -0.071], Standard Error of Mean 0.033

2. Secondary Outcome: Variability of Height SDS at 24 Months
Description: The continuous endpoint of variability of height SDS at 24 months was defined as the SD of the 24 month height SDS.
Time Frame: 2 years
Population: FAS included all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline height SDS value available. LOCF rule was applied to impute Month 24 missing height SDS data.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | Standard Dose Arm | Individualized Dose Arm
Number analyzed (Participants) | 114 | 202
Standard Deviation Score (SDS)
  Change from baseline at 24 months (n=101,184) | 1.12 (0.408) | 1.11 (0.518)
  Change from baseline at 24 months LOCF (n=114,202) | 1.03 (0.475) | 1.04 (0.544)
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm; Test type: Superiority or Other; p = 0.627, ANOVA (Levene's Test)

3. Secondary Outcome: Time Cost (Months Until >= -2 SDS)
Description: Time cost was defined as the number of months needed until height SDS was within the normal limit (ie, >= -2SDS).
Time Frame: 2 years
Population: Full analysis set (FAS) included all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline height SDS value available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Dose Arm | Individualized Dose Arm
Number analyzed (Participants) | 114 | 202
Months | 12.00 [8.00 to 12.00] | 12.00 [8.00 to 12.00]
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm; Test type: Superiority or Other; p = 0.8016, Regression, Cox; Hazard Ratio (HR) = 1.033, 95% CI 2-sided [0.802 to 1.330]

4. Secondary Outcome: Computed Cost of Height Gain at 48 Months
Description: The computed cost of height gain was defined as the amount of drug used relative to the observed height-gain, in terms of mg/cm, this was calculated at Month 48.
Time Frame: 4 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/cm
Groups:
- Individualized Dose Arm Overall: The participants received subcutaneous genotropin daily, at formula-calculated dose (up to maximum dose of 0.7 mg/kg/week) for the initial 2 years and then lowered to one of two approximately physiological doses (0.18 mg/kg/week or 0.24 mg/kg/week) for the remaining 2 years.
  The combined individualized dose group (N=202) includes 179 subjects who, at the start of the maintenance phase, were randomized to either 0.18 or 0.24 mg/kg/week dose subgroup. The remaining 23 subjects were not randomized at the start of the maintenance phase either due to early termination (n=19), or because they were initially randomized to the individualized dose, had the dose calculated to 0 mg, and had received the standard dose for the remainder of the study (n=4).
- Individualized Dose Arm 0.18 mg/kg/Week: The participants received subcutaneous genotropin daily, at formula-calculated dose (up to maximum dose of 0.7 mg/kg/week) for the initial 2 years and then lowered to one of two approximately physiological doses 0.18 mg/kg/week for the remaining 2 years.
- Individualized Dose Arm 0.24 mg/kg/Week: The participants received subcutaneous genotropin daily, at formula-calculated dose (up to maximum dose of 0.7 mg/kg/week) for the initial 2 years and then lowered to one of two approximately physiological doses 0.24 mg/kg/week for the remaining 2 years.
Arm/Group | Standard Dose Arm | Individualized Dose Arm Overall | Individualized Dose Arm 0.18 mg/kg/Week | Individualized Dose Arm 0.24 mg/kg/Week
Number analyzed (Participants) | 114 | 202 | 91 | 88
mg/cm | 72.77 (17.914) | 67.30 (24.382) | 63.07 (21.656) | 69.62 (21.903)
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm Overall; Test type: Superiority or Other; p = 0.0101, ANCOVA; Mean Difference (Final Values) = 5.822, 95% CI 2-sided [1.395 to 10.249], Standard Error of Mean 2.250
Statistical Analysis 2: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.18 mg/kg/Week; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 9.281, 95% CI 2-sided [4.417 to 14.145], Standard Error of Mean 2.471
Statistical Analysis 3: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.24 mg/kg/Week; Test type: Superiority or Other; p = 0.2001, ANCOVA; Mean Difference (Final Values) = 3.204, 95% CI 2-sided [-1.707 to 8.114], Standard Error of Mean 2.495

5. Secondary Outcome: Estimated Cost of Height Gain Estimated Until Full Adult Height (FAH) at 48 Months
Description: The estimated cost of long-term height gain until FAH was calculated.
Time Frame: 4 years
Population: Full analysis set (FAS) included all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline height SDS value available. LOCF rule was applied to impute Month 24 missing height SDS data.
Measure: Mean (Standard Deviation); unit: mg/cm
Groups:
- Individualized Dose Arm 0.24/mg/kg/Week: The participants received subcutaneous genotropin daily, at formula-calculated dose (up to maximum dose of 0.7 mg/kg/week) for the initial 2 years and then lowered to one of two approximately physiological doses 0.24 mg/kg/week for the remaining 2 years.
Arm/Group | Standard Dose Arm | Individualized Dose Arm Overall | Individualized Dose Arm 0.18 mg/kg/Week | Individualized Dose Arm 0.24/mg/kg/Week
Number analyzed (Participants) | 112 | 192 | 90 | 88
mg/cm | 127.99 (29.708) | 91.34 (31.854) | 80.06 (21.000) | 92.24 (25.213)
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm Overall; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 36.899, 95% CI 2-sided [30.181 to 43.618], Standard Error of Mean 3.414
Statistical Analysis 2: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.18 mg/kg/Week; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = 48.517, 95% CI 2-sided [42.054 to 54.980], Standard Error of Mean 3.284
Statistical Analysis 3: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.24/mg/kg/Week; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = 34.443, 95% CI 2-sided [27.936 to 40.951], Standard Error of Mean 3.306

6. Secondary Outcome: Change From Baseline in Height SDS at 48 Months.
Description: Change in height SDS was measured at 48 months.
Time Frame: 4 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | Standard Dose Arm | Individualized Dose Arm Overall | Individualized Dose Arm 0.18 mg/kg/Week | Individualized Dose Arm 0.24 mg/kg/Week
Number analyzed (Participants) | 114 | 202 | 91 | 88
Standard Deviation Score (SDS) | 1.33 (0.717) | 1.24 (0.668) | 1.33 (0.637) | 1.34 (0.633)
Statistical Analysis 1: Comparison: Standard Dose Arm vs Individualized Dose Arm Overall; Test type: Superiority or Other; p = 0.2618, ANCOVA; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.068 to 0.249], Standard Error of Mean 0.081
Statistical Analysis 2: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.18 mg/kg/Week; Test type: Superiority or Other; p = 0.8926, ANCOVA; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.172 to 0.198], Standard Error of Mean 0.094
Statistical Analysis 3: Comparison: Standard Dose Arm vs Individualized Dose Arm 0.24 mg/kg/Week; Test type: Superiority or Other; p = 0.9566, ANCOVA; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.192 to 0.181], Standard Error of Mean 0.095

ADVERSE EVENTS:
Time Frame: 4 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Standard Dose Arm | Individualized Dose Arm
Serious Adverse Events (participants affected / at risk) | 13/118 | 7/198
Other Adverse Events (participants affected / at risk) | 103/118 | 165/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Arm (N=118) | Individualized Dose Arm (N=198)
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Arm (N=118) | Individualized Dose Arm (N=198)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 19
Hypersensitivity (Immune system disorders) | 6 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 13
Headache (Nervous system disorders) | 33 | 59
Pyrexia (General disorders) | 13 | 22
Abdominal discomfort (Gastrointestinal disorders) | 2 | 10
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 9 | 17
Diarrhoea (Gastrointestinal disorders) | 7 | 12
Nausea (Gastrointestinal disorders) | 5 | 11
Vomiting (Gastrointestinal disorders) | 15 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 17
Scoliosis (Musculoskeletal and connective tissue disorders) | 11 | 19
Ear infection (Infections and infestations) | 1 | 11
Gastroenteritis (Infections and infestations) | 10 | 11
Gastroenteritis viral (Infections and infestations) | 7 | 15
Influenza (Infections and infestations) | 16 | 22
Nasopharyngitis (Infections and infestations) | 8 | 25
Otitis externa (Infections and infestations) | 2 | 10
Otitis media (Infections and infestations) | 11 | 23
Pharyngitis streptococcal (Infections and infestations) | 15 | 30
Sinusitis (Infections and infestations) | 9 | 23
Upper respiratory tract infection (Infections and infestations) | 28 | 45
Viral infection (Infections and infestations) | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.